CLINICAL TRIAL: NCT01143857
Title: Human Behavioral Pharmacology Laboratory Study of Varenicline's Impact on Cocaine Reinforcement
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Plebani (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Jennifer Plebani, Sponsor-Investigator, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 810580; K01DA025073 (NIH)
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Active Comparator)
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator)
  Interventions: Drug: Varenicline

INTERVENTIONS:
Drug: Varenicline — Varenicline 2.0 mg/day or Placebo

SUMMARY:
Cocaine use, abuse and dependence is a public health problem that is directly responsible for hundreds of billions of dollars in health care expenditures per year. Relapse rates to cocaine use are high, creating a pressing need to develop effective therapies for cocaine dependence. The proposed research will focus on investigating the determinants and consequences of cocaine dependence via measurement of physiological, behavioral and subjective effects of acute doses of cocaine in healthy non-drug dependent human volunteers in the laboratory, and through examination of the effects of pharmacotherapies on the above effects of cocaine. This study will examine cocaine-derived reinforcement under week-long sub-chronic varenicline (Chantix) dosing, and under placebo conditions. The study is a within-subjects crossover design using 24 subjects. Subjects will be screened and consented into the study at the Treatment Research Center (TRC). Study visits where behavioral and physiological outcome data will be obtained will be conducted at the Clinical and Translational Research Center (CTRC) of the Hospital of the University of Pennsylvania. Subjects will be outpatients for this trial, with CTRC sessions scheduled at least one week apart.

ELIGIBILITY:
Inclusion Criteria

1. Males and females, 18 to 60 years old.
2. Recreational users of cocaine reporting at least six instances of cocaine use in the past 12 months and at least one use in the past 30 days.
3. Live within a commutable distance of the Treatment Research Center (TRC) at the Penn/VA Center for Studies of Addiction, University of Pennsylvania. We define this to be a distance within the service area of Septa, within an hour drive, or a distance that both the patient and Principal Investigator (PI) find acceptable.
4. Understands and signs the informed consent.

Exclusion Criteria:

1. Current DSM-IV diagnosis of any psychoactive substance dependence other than nicotine dependence, as determined by the Structured Clinical Interview for the DSM (SCID).
2. Current severe psychiatric symptoms (e.g., psychosis, dementia, suicidal or homicidal ideation, mania or depression requiring anti-depressant therapy) as diagnosed using the SCID, the Hamilton Anxiety Rating Scale (Ham A), and Hamilton Ration Scale for Depression (HAM-D).
3. Individuals scoring > 10 on the Hamilton Rating Scale for Depression (HAM-D).
4. Use of any investigational medication within the past 30 days.
5. Concomitant treatment with psychotropic medications.
6. Concomitant use of any one of the following drugs or classes of drugs:

   * Reserpine
   * Verapamil
   * theophylline,
   * trimethoprim,
   * cimetidine,
   * haloperidol,
   * benzodiazepines, or
   * antiepileptic drugs (AEDs).
7. Patients with a known hypersensitivity to varenicline.
8. Patients with severe concurrent illnesses such as bronchospastic disease, hyperthyroidism, diabetes mellitus.
9. Patients with known AIDS or other serious illnesses that may require hospitalization during the study.
10. Female subjects who are pregnant or lactating, or female subjects of child-bearing potential who are not using acceptable methods of birth control; acceptable methods of birth control include:

    * Barrier method (diaphragm or condom) with spermicide
    * Intrauterine progesterone contraceptive system
    * Levonorgesterel implant
    * Medroxyprogesterone acetate contraceptive injection, or
    * Oral contraceptives.
11. Patients with impaired renal function, as indicated by corrected creatinine clearance below 60 ml/min/70 kg as determined by the modified Cockcroft equation (CDC, 1986).
12. An unacceptable liver panel (liver function tests; LFTs) that may be indicative of hepatic dysfunction.
13. Clinical laboratory tests (e.g., CBC, blood chemistries, urinalysis) outside normal limits.
14. History of significant heart disease or dysfunction (e.g., an arrhythmia which required medication, Wolff Parkinson -White Syndrome, angina pectoris, documented history of myocardial infarction, heart failure).
15. Electrocardiography (EKG) indicative of 1st degree heart block, sinus tachycardia, left-axis deviation, non-specific ST or T-wave changes.
16. History of chest pain associated with cocaine use that prompted a visit to a physician.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Varenicline's impact on reinforcing effects of cocaine | 6 weeks
  The primary aim of this study is to examine what impact sub-chronic dosing with varenicline has on the subjective and reinforcing effects of cocaine and on cocaine self-administration in cocaine experienced individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Treatment Research Center, Philadelphia, Pennsylvania, United States